CLINICAL TRIAL: NCT03357614
Title: Prospective, Phase 3, Randomized, Multi-center, Double-blind, Double-dummy Study of Efficacy, Tolerability & Safety of Sulopenem Followed by Sulopenem-etzadroxil/Probenecid vs Ertapenem Followed by Cipro for Treatment of cUTI in Adults
Brief Title: Sulopenem Followed by Sulopenem-etzadroxil/Probenecid vs Ertapenem Followed by Cipro for Complicated UTI in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT001-302
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2019-11

CONDITIONS: Complicated Urinary Tract Infections
MeSH Terms: interventions — sulopenem; Probenecid; Ertapenem; Ciprofloxacin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulopenem (Experimental): Sulopenem 1000 mg IV once daily for a minimum of 5 days, followed by sulopenem-etzadroxil/probenecid 500 mg PO twice daily to complete 7-10 total days of treatment
  Interventions: Drug: Sulopenem; Drug: Sulopenem-Etzadroxil/Probenecid
- Ertapenem (Active Comparator): Ertapenem 1000 mg IV once daily for a minimum of 5 days, followed by ciprofloxacin 500 mg PO twice daily or amoxicillin-clavulanate 500 mg PO twice daily to complete 7-10 total days of treatment
  Interventions: Drug: Ertapenem; Drug: Ciprofloxacin; Drug: Amoxicillin-clavulanate

INTERVENTIONS:
Drug: Sulopenem — Antibiotic therapy for complicated UTI
  Arms: Sulopenem
Drug: Sulopenem-Etzadroxil/Probenecid — Antibiotic therapy for complicated UTI
  Arms: Sulopenem
Drug: Ertapenem — Antibiotic therapy for complicated UTI
  Other Names: Invanz
  Arms: Ertapenem
Drug: Ciprofloxacin — Antibiotic therapy for complicated UTI
  Other Names: Cipro
  Arms: Ertapenem
Drug: Amoxicillin-clavulanate — Antibiotic therapy for complicated UTI
  Other Names: Augmentin
  Arms: Ertapenem

SUMMARY:
This is a prospective, phase 3, randomized, multicenter, double-blind, double-dummy study to compare the efficacy and safety of sulopenem followed by sulopenem-etzadroxil/probenecid versus ertapenem followed by ciprofloxacin for the treatment of complicated urinary tract infections (cUTI) in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age with more than 24 hours of urinary symptoms attributable to a UTI
2. Able to provide informed consent
3. Clinically documented pyelonephritis or complicated urinary tract infection:

   1. Pyelonephritis with normal anatomy
   2. Complicated UTI as defined by one or more of the following factors:

   i. The presence of an indwelling catheter ii. >100 mL of residual urine after voiding iii. Neurogenic bladder iv. Obstructive uropathy due to nephrolithiasis, tumor or fibrosis v. Azotemia due to intrinsic renal disease vi. Urinary retention in men possibly due to benign prostatic hypertrophy vii. Surgically modified or abnormal urinary tract anatomy
4. At least two of the following signs or symptoms:

   1. Rigors, chills or fever/hypothermia
   2. Flank pain or pelvic pain
   3. Nausea or vomiting
   4. Dysuria, urinary frequency or urinary urgency
   5. Costovertebral angle tenderness on physical examination
5. A mid-stream urine specimen with:

   1. a dipstick analysis positive for nitrite AND
   2. evidence of pyuria as defined by either: i. a dipstick analysis positive for leukocyte esterase AND/OR ii. at least 10 white blood cells per cubic millimeter on microscopic analysis of unspun urine AND/OR iii. White blood cell count ≥10 cells/high-powered field in urine sediment

Exclusion Criteria

1. Receipt of effective antibacterial drug therapy for complicated urinary tract infection (cUTI) for a continuous duration of more than 24 hours during the previous 72 hours. Patients who have objective documentation of clinical progression of cUTI while on antibacterial drug therapy, or patients who received antibacterial drugs for surgical prophylaxis and then develop cUTI, may be appropriate for enrollment.
2. Subjects with an organism isolated from the urine within the last year known to be resistant to ertapenem
3. Severe structural or functional urinary tract abnormality responsible for an intractable infection which in the opinion of the investigator would require > 10 days of therapy or post-treatment prophylaxis (eg. patients with chronic vesiculo-ureteral reflux).
4. Uncomplicated UTI
5. Patients with paraplegia/quadriplegia
6. Hypotension with systolic blood pressure < 90 mm Hg
7. Complicated UTI associated with complete obstruction, emphysematous pyelonephritis, known or suspected renal or perinephric abscess or expected to require surgical intervention (not placement of catheters) to achieve cure
8. Patients with a known history of myasthenia gravis
9. Patients who require concomitant administration of tizanidine or valproic acid
10. Patients with a history of allergy to carbapenems or quinolones or amoxicillin-clavulanate or other beta-lactams, or hypersensitivity to probenecid
11. Renal transplantation
12. Patients requiring dialysis
13. Acute or chronic prostatitis
14. High risk for cUTI caused by Pseudomonas sp. (eg,. history of prior UTI due to Pseudomonas species, recent steroid use, others)
15. Chronic indwelling catheters or stents
16. Ileal loops or vesico-urethral reflux
17. Recent trauma to the pelvis or urinary tract within the prior 30 days
18. History of seizures
19. Patients with a history of blood dyscrasias
20. Patients with a history of uric acid kidney stones
21. Patients with acute gouty attack
22. Patients on chronic methotrexate therapy
23. Females of child-bearing potential who are unable to take adequate contraceptive precautions, have a positive pregnancy test result within 24 hours of study entry, are otherwise known to be pregnant, or are currently breastfeeding an infant.
24. Male subjects must agree to use of an effective barrier method of contraception during the study and for 14 days post treatment
25. Patients known to have a history of liver or kidney disease or neutropenia as defined by the following baseline laboratory criteria:

    * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 3 X Upper Limit of Normal
    * Total bilirubin > 2 X Upper Limit of Normal
    * Neutropenia (<1000 cells/mm3)
26. Patients participating in any other clinical study that involved the administration of an investigational medication
27. Patient immunocompromised
28. Patients unlikely to comply with the protocol
29. Patients considered unlikely to survive the 4-week study period or has a rapidly progressive or terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (14):
  - Medical Facility, Bellflower, California
  - Medical Facility, Chula Vista, California
  - Medical Facility, La Mesa, California
  - Medical Facility, La Palma, California
  - Medical Facility, Torrance, California
  - Medical Facility, Miami Lakes, Florida
  - Medical Facility, Columbus, Georgia
  - Medical Facility, Idaho Falls, Idaho
  - Medical Facility, Boston, Massachusetts
  - Medical Facility, Royal Oak, Michigan
  - Medical Facility, Butte, Montana
  - Medical Facility, Columbus, Ohio
  - Medical Facility, Dallas, Texas
  - Medical Facility, Houston, Texas
- Estonia (3):
  - Medical Facility, Kohtla-Järve
  - Medical Facility, Tallinn
  - Medical Facility, Võru
- Medical Facility, Tbilisi, Georgia
- Hungary (6):
  - Medical Facility, Baja
  - Medical Facility, Budapest
  - Medical Facility, Nagykanizsa
  - Medical Facility, Nyíregyháza
  - Medical Facility, Szentes
  - Medical Facility, Tatabánya
- Latvia (4):
  - Medical Facility, Daugavpils
  - Medical Facility, Liepāja
  - Medical Facility, Riga
  - Medical Facility, Valmiera

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunne MW, Aronin SI, Das AF, Akinapelli K, Breen J, Zelasky MT, Puttagunta S. Sulopenem for the Treatment of Complicated Urinary Tract Infections Including Pyelonephritis: A Phase 3, Randomized Trial. Clin Infect Dis. 2023 Jan 6;76(1):78-88. doi: 10.1093/cid/ciac704. PMID 36068705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sulopenem | Ertapenem
Started | 697 | 698
Completed | 672 | 670
Not Completed | 25 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulopenem | Ertapenem | Total
Number analyzed (Participants) | 697 | 698 | 1395
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (18.2) | 59.3 (18.2) | 58.5 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 389 | 380 | 769
  Male | 308 | 318 | 626
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 42
  Not Hispanic or Latino | 672 | 675 | 1347
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Latvia | 31 | 42 | 73
  Hungary | 70 | 47 | 117
  United States | 30 | 31 | 61
  Georgia | 81 | 92 | 173
  Estonia | 16 | 18 | 34
  Bulgaria | 150 | 145 | 295
  Czechia | 8 | 10 | 18
  Poland | 3 | 3 | 6
  Russia | 180 | 194 | 374
  Serbia | 1 | 4 | 5
  Slovakia | 10 | 8 | 18
  Ukraine | 109 | 98 | 207
  Croatia | 8 | 6 | 14
Diabetes [Count of Participants; unit: Participants] | 114 | 114 | 228

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Success
Description: Clinical success is defined as complete resolution of cUTI symptoms present at study entry and no new cUTI symptoms; microbiologic success is defined as eradication of the bacterial pathogen found at study entry (reduced to <1000 CFU/mL)
Time Frame: Day 21 +/- 1 day
Population: Analysis population is the microbiologic modified intent-to-treat population (all modified intent-to-treat patients with a positive study entry urine culture within 48 hours prior to first dose, defined as >100,000 CFU/mL of a uropathogen and no more than 2 species of a uropathogen >100,000 CFU/mL; if 1 of the uropathogens was also isolated from baseline blood culture, however, the patient was included in this population regardless of the baseline urine culture result).
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem | Ertapenem
Number analyzed (Participants) | 444 | 440
Participants | 301 | 325

2. Secondary Outcome: Percentage of Participants With Microbiologic Success
Description: Microbiologic success is defined as demonstrating <1000 CFU/mL of the baseline urpathogen by quantitative urine culture
Time Frame: Day 21 +/- 1 day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem | Ertapenem
Number analyzed (Participants) | 444 | 440
Participants | 316 | 343

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the final visit, an average of 28 days.
Arm/Group | Sulopenem | Ertapenem
All-Cause Mortality (participants affected / at risk) | 2/697 | 0/698
Serious Adverse Events (participants affected / at risk) | 14/697 | 6/698
Other Adverse Events (participants affected / at risk) | 0/697 | 0/698
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem (N=697) | Ertapenem (N=698)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs will provide Iterum opportunity to review proposed publication/other type of disclosure before it's submitted/otherwise disclosed. PI will provide manuscripts, abstracts, or full text of intended disclosure (poster, invited speaker presentation, etc) to Iterum at least 30 days before submitted for publication/otherwise disclosed. If any patent action is required to protect intellectual property rights, PI agrees to delay disclosure for a period not to exceed an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT03357614/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03357614/SAP_001.pdf